CLINICAL TRIAL: NCT06365840
Title: PHASE 2 STUDY OF IMC-001 IN PATIENTS WITH METASTATIC OR LOCALLY ADVANCED TMB-H SOLID TUMOR
Brief Title: A Study of IMC-001 In Patients With Metastatic Or Locally Advanced TMB-H Solid Tumor
Acronym: TMB-H
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ImmuneOncia Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMC-001-202
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: TMB-H; Histologically or Cytologically Proven Metastatic or Locally Advanced Solid Tumors
Keywords: IMC-001,IMC-001-202,TMB-H
MeSH Terms: interventions — IMC-001

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMC-001 (Experimental)
  Interventions: Drug: IMC-001

INTERVENTIONS:
Drug: IMC-001 — All participants will receive the study drug, IMC-001, at 20 mg/kg Q2W via IV infusion over 60 minutes.

SUMMARY:
The goal of this clinical trial is to determine the efficacy of IMC-001 in metastatic or locally advanced TMB-H solid tumor patients.

ELIGIBILITY:
Inclusion Criteria:

1. Documented TMB-H:≥ 16 mut/Mb, determined by the TruSightTM Oncology 500 NGS panel or OncomineTM Comprehensive Assay Plus
2. Histologically or cytologically proven metastatic or locally advanced solid tumors.The participant must have at least one measurable tumor lesion per RECIST 1.1.
3. Investigator has confirmation that participant's tumor tissue is available to be submitted to a central pathology laboratory.
4. Adult age(as defined by respective country)
5. The nature of the study and voluntarily sign an ICF
6. ECOG 0 or1
7. Prior systemic radiation therapy must be completed at least 4 weeks before the first dose of study drug. Prior focal radiotherapy must be completed at least 2 weeks before the first dose of study drug.
8. At the time of the first dose of study drug at least 28 days since the last chemotherapy, immunotherapy, biological or investigational therapy, and have recovered from toxicities associated with such treatment to < Grade 2.
9. Adequate hematologic function, hepatic function, and renal function
10. Female participants must meet one of the following criteria:

    * Postmenopausal (≥24 months, or ≥12 months with FSH > 40 IU/L),
    * surgically incapable of bearing children (i.e., has had a hysterectomy or bilateral oophorectomy); or
    * females of childbearing potential must agree to use a reliable form of contraceptive during the study treatment period and for at least 90 days following the last dose of study drug.
11. Male participants must agree to use barrier contraception (i.e., condoms) for the duration of the study and for at least 90 days after the last dose of study drug.
12. Predicted life expectancy of at least 16 weeks.

Exclusion Criteria:

1. Previously treated with an anti-PD-L1 or anti-PD-1 antibody
2. Known presence of symptomatic CNS metastases
3. Any active autoimmune disease or a documented history of autoimmune disease
4. Apparent active and known viral infection with HIV, hepatitis B virus or hepatitis C virus
5. Pregnant or lactating

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
ORR | Imaging every 6 weeks (±7 days) until PD or other anticancer therapy, during treatment (including EOT visit) and follow-up. EOT: 28 days (±3) after last dose. Max treatment: 2 years (52 cycles, each cycle is 14 days).
  Percentage of participants achieving a best overall response (BOR) of CR or PR by centralized independent review using RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Evaluate additional efficacy variables of IMC-001 | through study completion, an average of 1 year
  Terms, frequency, severity, and seriousness of adverse events (AEs) and relationship of AEs to IMC-001
Evaluate additional efficacy variables of IMC-001 : Progression-Free Survival (PFS) | Imaging every 6 weeks (±7 days) until PD or other anticancer therapy, during treatment (including EOT visit) and follow-up. EOT: 28 days (±3) after last dose. Max treatment: 2 years (52 cycles, each cycle is 14 days).
  Progression-Free Survival (PFS), (Unit of Measure: Months) Variables determined by the centralized independent assessment and Investigator's assessment based on RECIST Version 1.1
Evaluate additional efficacy variables of IMC-001 : Duration of Response (DOR) | Imaging every 6 weeks (±7 days) until PD or other anticancer therapy, during treatment (including EOT visit) and follow-up. EOT: 28 days (±3) after last dose. Max treatment: 2 years (52 cycles, each cycle is 14 days).
  Duration of Response (DOR), (Unit of Measure: Months) Variables determined by the centralized independent assessment and Investigator's assessment based on RECIST Version 1.1
Evaluate additional efficacy variables of IMC-001 : Time to Progression (TTP) | Imaging every 6 weeks (±7 days) until PD or other anticancer therapy, during treatment (including EOT visit) and follow-up. EOT: 28 days (±3) after last dose. Max treatment: 2 years (52 cycles, each cycle is 14 days).
  Time to Progression (TTP), (Unit of Measure: Months) Variables determined by the centralized independent assessment and Investigator's assessment based on RECIST Version 1.1
Evaluate additional efficacy variables of IMC-001 : Disease Control Rate (DCR) | Imaging every 6 weeks (±7 days) until PD or other anticancer therapy, during treatment (including EOT visit) and follow-up. EOT: 28 days (±3) after last dose. Max treatment: 2 years (52 cycles, each cycle is 14 days).
  Disease Control Rate (DCR), (Unit of Measure: Percentage of participants) Variables determined by the centralized independent assessment and Investigator's assessment based on RECIST Version 1.1
Evaluate additional efficacy variables of IMC-001 : Objective Response Rate (ORR) | Imaging every 6 weeks (±7 days) until PD or other anticancer therapy, during treatment (including EOT visit) and follow-up. EOT: 28 days (±3) after last dose. Max treatment: 2 years (52 cycles, each cycle is 14 days).
  Objective Response Rate (ORR), (Unit of Measure: Percentage of participants) Variables determined by the Investigator's assessment based on RECIST Version 1.1
Evaluate additional efficacy variables of IMC-001 : Immune progression-free survival (iPFS) | Imaging every 6 weeks (±7 days) until PD or other anticancer therapy, during treatment (including EOT visit) and follow-up. EOT: 28 days (±3) after last dose. Max treatment: 2 years (52 cycles, each cycle is 14 days).
  Immune progression-free survival (iPFS), (Unit of Measure: Months) Variables determined by the centralized independent assessment and Investigator's assessment based on immune RECIST (iRECIST)
Evaluate additional efficacy variables of IMC-001 : Immune duration of response (iDOR) | Imaging every 6 weeks (±7 days) until PD or other anticancer therapy, during treatment (including EOT visit) and follow-up. EOT: 28 days (±3) after last dose. Max treatment: 2 years (52 cycles, each cycle is 14 days).
  Immune duration of response (iDOR), (Unit of Measure: Months) Variables determined by the centralized independent assessment and Investigator's assessment based on immune RECIST (iRECIST)
Evaluate additional efficacy variables of IMC-001 : Immune objective response rate (iORR) | Imaging every 6 weeks (±7 days) until PD or other anticancer therapy, during treatment (including EOT visit) and follow-up. EOT: 28 days (±3) after last dose. Max treatment: 2 years (52 cycles, each cycle is 14 days).
  Immune objective response rate (iORR), (Unit of Measure: Percentage of participants) Variables determined by the centralized independent assessment and Investigator's assessment based on immune RECIST (iRECIST)
Survival Outcome : Overall Survival (OS) | through study completion, an average of 1 year
  Overall Survival (OS), (Unit of Measure: Months)
Evaluate the pharmacokinetic (PK) profile of IMC-001 | through study completion, an average of 1 year
  IMC-001 PK parameter: observed serum concentration immediately before dosing (Ctrough)
Characterize the immunogenicity of IMC-001 | through study completion, an average of 1 year
  Incidence of anti-drug antibody and neutralizing antibody (NAb) (including serum titers of anti-IMC-001 antibodies)

CONTACTS AND LOCATIONS:
Overall Officials: JEEYUN LEE, Principal Investigator — Samsung Medical Center, Republic of Korea
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No